CLINICAL TRIAL: NCT04133233
Title: Low Dose IL-2 Therapy in Patients With a Depressive Episode in the Course of a Bipolar Disorder
Acronym: DEPIL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D20180617; 2018-002777-22 (EudraCT Number); MEDAECNAT-2018-10-00069 (Other: ANSM)
Record Dates: First submitted 2019-09-17; First posted 2019-10-21 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Depression
Keywords: Low dose of IL-2; Treg response
MeSH Terms: conditions — Bipolar Disorder | interventions — Interleukin-2

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled (2 active: 1 placebo), multicentre, 6-week, proof-of concept trial of add on low dose IL-2 therapy in patients with a depressive episode in the course of a bipolar disorder, hospitalized or not. The study will be an add-on study, with no wash-out period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active treatment (Experimental): IL-2 (ILT-101) Sub-cutaneous
  1 million UI/j
  Interventions: Drug: ILT101
- placebo (Placebo Comparator): placebo Sub-cutaneous The Placebo used is a sterile powder that will be produced by the CMO (AMATSI, France).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: ILT101 — Treatment administration consists in a first course of five-day treatment (induction), followed by a single injection every week for 4 weeks (maintenance; from Week 3 to Week 6)
  Other Names: IL2
  Arms: active treatment
Drug: Placebos — Treatment administration consists in a first course of five-day treatment (induction), followed by a single injection every week for 4 weeks (maintenance; from Week 3 to Week 6)
  Other Names: placebo
  Arms: placebo

SUMMARY:
The purpose of this study will be to demonstrate improvement of the T regulatory cells (Treg) response, under add on low-dose Interleukin 2 (ld-IL2) in patients with bipolar disorders experiencing a depressive relapse

DETAILED DESCRIPTION:
A hypothesis still under study concerning the pathophysiological mechanisms of bipolar disorder concerns an immunological disorder that could possibly be involved in this disease and during a depressive episode. In particular, that the multiplication of a certain category of white blood cells called "regulators" that block the toxic effect of more aggressive white blood cells could improve these disorders.

The aim of this research is therefore to check the effectiveness and safety of injections of Interleukin 2 (IL-2) to induce this multiplication of regulatory white blood cells.

IL-2 is a natural protein released by white blood cells that is used for the proper functioning of the immune defence system. The favourable effects of injecting small doses of IL-2 are known and assessed in other diseases, including autoimmune diseases.

The secondary objective of this study is to assess the effect of these injections on patient's mood, which could be improved by this treatment.

ELIGIBILITY:
Inclusion Criteria:

* A depressive episode according to DSM-V criteria in the course of a bipolar disorder
* MADRS score > 17
* Already on a mood stabilizer and/or antidepressant
* Patient with a normal or controlled thyroid function
* Male or female both using effective methods of contraception during treatment if sexually active.

Exclusion Criteria:

* - Contraindication to IL-101 therapy:
* Hypersensitivity to active substance or excipient;
* Active infection requiring antibiotics therapy;
* Organ failure (e.g., liver, kidney, lung and heart);
* Immunosuppressed patient
* Hepatotoxic, nephrotoxic, myelotoxic or cardiotoxic drugs
* Other chronic diseases
* Signs of active infection requiring treatment
* Previous history of organ transplantation
* Leukocytes < 4000 / mm3, platelets < 100 000 / mm3, Hemoglobin < 10.0 g/dL or 6.2 mmol/L, red cell blood < 3.5 T/L.
* Anti-TPO or anti-TG or anti-TRACKS positive at inclusion.
* Use of anti-inflammatory medication on a regular basis for a chronic inflammatory/autoimmune Disorder (NSAD, immunosuppressant IV-Ig based treatment);
* Ongoing fever < 38
* uncontrolled diabetes type I or II;
* Existing cancer or history of cancer in the last 5 years (except skin epidermoid cancer or in-situ cervix cancer);
* Existing or planned pregnancy or lactation;
* Person under legal protection (1121-8 of CSP, Public Health Code
* Pregnant and parturient and Breast feeding women (1121-5 of CSP)
* legally detained person (1121-6 of CSP)
* hospitalisation without consent
* under the age of majority (1121-7of CSP)
* Immediate risk for suicidal behaviour (MADRS-item 10 >2 or columbia > 2 for suicide idea);
* Known HIV infection or clinically manifest Acquired Immune Deficiency Syndrome (AIDS), Parkinson's or Alzheimer's disease, or any other serious condition likely to interfere with the conduct of the trial;
* Participation to an interventional study concomitantly or within 30 days prior to this study, except in the cohorts studies aiming at the analysis of immuno-inflammatory biomarkers and/or brain imaging studies.
* Patients thought to be unreliable or incapable of complying with the requirements of the protocol;
* Patient is relative of, or staff directly reporting to the investigator;
* Patient is employee of the sponsor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
change of Treg response | baseline to Day 5
  Percentage Treg fold increase compared to baseline at Day 5

SECONDARY OUTCOMES:
Treg response, under ld-IL2 in relation with symptomatic assessment of mood improvements | from baseline to week 6
  Change in the value of Montgomery Asberg Depression Rating and in The inventory of depressive symptomatology
changes in immune homeostasis under ld-IL2 in relation with symptomatic assessment of mood improvements | between Day 5 and Day 60
  variation in Treg /CD4+ at different visit expressed as percentage of baseline value
Assess the incidence of ld-IL2(safety and tolerability) in patients with a depressive episode in the course of a bipolar disorder | baseline to Day 60
  Frequency and type of adverse events during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Leboyer, Pr, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pr Marion Leboyer, Créteil, Hôpital Albert Chenevier, France

REFERENCES:
- [Derived] Leboyer M, Foiselle M, Tchitchek N, Tamouza R, Lorenzon R, Richard JR, Arrouasse R, Le Corvoisier P, Le Dudal K, Vicaut E, Ellul P, Rosenzwajg M, Klatzmann D. Low-dose interleukin-2 in patients with bipolar depression: A phase 2 randomised double-blind placebo-controlled trial. Brain Behav Immun. 2025 Jan;123:177-184. doi: 10.1016/j.bbi.2024.09.005. Epub 2024 Sep 4. PMID 39242054
- [Derived] Poletti S, Zanardi R, Mandelli A, Aggio V, Finardi A, Lorenzi C, Borsellino G, Carminati M, Manfredi E, Tomasi E, Spadini S, Colombo C, Drexhage HA, Furlan R, Benedetti F. Low-dose interleukin 2 antidepressant potentiation in unipolar and bipolar depression: Safety, efficacy, and immunological biomarkers. Brain Behav Immun. 2024 May;118:52-68. doi: 10.1016/j.bbi.2024.02.019. Epub 2024 Feb 15. PMID 38367846